CLINICAL TRIAL: NCT05325541
Title: Effects of Visual Biofeedback Therapy on Balance, Freezing of Gait and Cognition Among Stage III Parkinson's Patients: A Randomized Controlled Trial
Brief Title: Effects of Visual Biofeedback Therapy in Parkinson's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4471121FHREH
Record Dates: First submitted 2022-03-22; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Experimental: Game-Based Rehabilitation: Device: Visual Biofeedback Therapy Session Visual Biofeedback intervention will be given for 24 sessions, comprising of 45-50 minutes, 3 times/week for the duration of 8 weeks.
  Placebo Comparator: Conventional Rehabilitation: Conventional Balance exercise Conventional Balance exercises will be given for 24 sessions, comprising of 45-50 minutes, 3 times/week for the duration of 8 weeks.
Who Masked: Participant
Masking Description: All participants will be blinded regarding treatment. A total of 36 patients will be recruited and assigned into two groups. Group A will receive visual biofeedback balance exercises and Group B will receive Conventional balance exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms 1 (Experimental): Game-Based Rehabilitation received total 24 sessions, 45-50 minutes/session, 3 times/week for total 8 weeks.
  Interventions: Device: Visual Biofeedback Therapy
- Arms 2 (Placebo Comparator): Conventional Rehabilitation received total 24 sessions, 45-50 minutes/session, 3 times/week for total 8 weeks.
  Interventions: Behavioral: Conventional Balance exercise

INTERVENTIONS:
Device: Visual Biofeedback Therapy — Visual Biofeedback intervention will be given for 24 sessions, comprising of 45-50 minutes, 3 times/week for the duration of 8 weeks.
  Arms: Arms 1
Behavioral: Conventional Balance exercise — Conventional Balance exercises will be given for 24 sessions, comprising of 45-50 minutes, 3 times/week for the duration of 8 weeks.
  Arms: Arms 2

SUMMARY:
Parkinson's disease (PD) affects approximately 6.5 million people around the world and it is ranked as the second most common age-related neurodegenerative disease after Alzheimer disease. US have reported 800,000 PD patients in 2016, the highest number of reported PD patients in the world while UK has the lowest number of PD cases i.e. 100,000. With a rise of 2.3 million cases in 2026, an approximate annual growth rate of 2.52% is predicted globally. According to Pakistan Parkinson's society, approximately 450,000 Pakistanis were affected with PD. The age-specific prevalence of PD in Pakistan was found to be high in 70 to 79 years of age with males being more affected as compared to females. Parkinson's disease is a neurological condition, characterized by tremors, rigidity, and stiffness in the body, along with bradykinesia, walking and balance problems. Poor balance is one of the major and most disabling characteristics among Parkinson patients. Freezing of gait (FOG) and postural instability is one of the major cause of fall and loss of independence among PD patients whereas cognitive dysfunction is one of the common non-motor symptoms affecting 20 to 57% of PD patients. Among recent technological advancements in neurological physical therapy, virtual reality (VR) games have become an area of interest for researchers. Despite advances in the rehabilitation of PD, evidence regarding the effects of visual biofeedback therapy on Parkinson patients is still scarce. Only few studies have studied the effects of visual biofeedback therapy on balance in PD patients, but as per knowledge of the researcher there is no study published on effects of visual biofeedback therapy on FOG and cognition among Parkinson patients in Pakistan. Therefore, the present study is aimed to assess the effects of biofeedback balance training using a balance board on balance, FOG and cognition in patients with Parkinson disease.

DETAILED DESCRIPTION:
A total number of 36 patients will be recruited in the study. After the voluntary consent, all the patients will be randomly divided into Group A and B through the envelope method of simple random sampling. In addition, a total of 36 sealed envelopes, comprised of 18 envelopes for each group will be presented to the patients. Each patient will be asked to select one envelope of their choice. Upon selection of the envelope, patients will be allocated to the respective group. Thus, each group will comprise 18 patients respectively. Afterward, pre-assessment will be performed for each patient on all three outcome measures i.e. FRT, FOG-Q, and MoCA. A total of 36 patients will be recruited and assigned into two groups. Group A will receive visual biofeedback balance exercises and Group B will receive Conventional balance exercises. The intervention will be given for 8 consecutive weeks to each group. The training session will be based on a warm-up session for 5 to 10 minutes to each group followed by 30 minutes' session of visual biofeedback therapy for group A and 30 minutes balance exercises for group B and a cool-down period of 5 to 10 minutes excluding intervals of 1-minute rest after 5 minutes of activity. A trial will be terminated, if the patient reported ataxia, vertigo and syncope, feeling of fatigue and difficulty during exercise through fatigue severity scale and subjects unwilling to perform exercise.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease of age between 60-79 years.
* Diagnosed PD stage III.

Exclusion Criteria:

* Other neurological problems (Multiple sclerosis, amyotrophic lateral sclerosis and myasthenia gravis).
* Migraine.
* Auditory or visual deficits.
* Orthostatic hypotension.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Balance | Baseline
  Balance function will be assessed through Functional Reach Test FRT among stage III PD patients where high values indicates increase in balance function
Balance | After 8 weeks
  Balance function will be assessed through Functional Reach Test FRT among stage III PD patients where high values indicates increase in balance function
Freezing of Gait (FOG) | Pre-Treatment
  Freezing of Gait will be assessed through FOG Questionnaire among stage III PD patients where low values indicates decrease in freezing of gait
Freezing of Gait (FOG) | After 8 weeks
  Freezing of Gait will be assessed through FOG Questionnaire among stage III PD patients where low values indicates decrease in freezing of gait
Cognitive Function | Pre-Treatment
  Cognitive Function will be assessed using Montreal Cognitive Assessment among stage III PD patients where high values indicates increase in Cognitive Function
Cognitive Function | After 8 weeks
  Cognitive Function will be assessed using Montreal Cognitive Assessment among stage III PD patients where high values indicates increase in Cognitive Function

CONTACTS AND LOCATIONS:
Overall Officials: Fouzia Hussain, MPhil, Principal Investigator — Ziauddin University Karachi, Sindh, Pakistan
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilar-Navarro SG, Mimenza-Alvarado AJ, Palacios-Garcia AA, Samudio-Cruz A, Gutierrez-Gutierrez LA, Avila-Funes JA. Validity and Reliability of the Spanish Version of the Montreal Cognitive Assessment (MoCA) for the Detection of Cognitive Impairment in Mexico. Rev Colomb Psiquiatr (Engl Ed). 2018 Oct-Dec;47(4):237-243. doi: 10.1016/j.rcp.2017.05.003. Epub 2017 Jul 29. English, Spanish. PMID 30286846
- [Background] Feng YS, Yang SD, Tan ZX, Wang MM, Xing Y, Dong F, Zhang F. The benefits and mechanisms of exercise training for Parkinson's disease. Life Sci. 2020 Mar 15;245:117345. doi: 10.1016/j.lfs.2020.117345. Epub 2020 Jan 22. PMID 31981631
- [Background] Ferraz DD, Trippo KV, Duarte GP, Neto MG, Bernardes Santos KO, Filho JO. The Effects of Functional Training, Bicycle Exercise, and Exergaming on Walking Capacity of Elderly Patients With Parkinson Disease: A Pilot Randomized Controlled Single-blinded Trial. Arch Phys Med Rehabil. 2018 May;99(5):826-833. doi: 10.1016/j.apmr.2017.12.014. Epub 2018 Jan 11. PMID 29337023
- [Background] Gupta DK, Fahn S, Tatsuoka C, Kang UJ. Hoehn and Yahr stage 3 and postural stability item in the movement disorder society-unified Parkinson's disease rating scale. Mov Disord. 2018 Jul;33(7):1188-1189. doi: 10.1002/mds.27453. No abstract available. PMID 30153396
- [Background] Hulzinga F, Nieuwboer A, Dijkstra BW, Mancini M, Strouwen C, Bloem BR, Ginis P. The New Freezing of Gait Questionnaire: Unsuitable as an Outcome in Clinical Trials? Mov Disord Clin Pract. 2020 Jan 14;7(2):199-205. doi: 10.1002/mdc3.12893. eCollection 2020 Feb. PMID 32071940
- [Background] Khan S, Nabi G, Naeem M, Ali L, Silburn PA, Mellick GD. A door-to-door survey to estimate the prevalence of Parkinsonism in Pakistan. Neuropsychiatr Dis Treat. 2016 Jun 21;12:1499-506. doi: 10.2147/NDT.S86329. eCollection 2016. PMID 27382292
- [Background] Negrini S, Bissolotti L, Ferraris A, Noro F, Bishop MD, Villafane JH. Nintendo Wii Fit for balance rehabilitation in patients with Parkinson's disease: A comparative study. J Bodyw Mov Ther. 2017 Jan;21(1):117-123. doi: 10.1016/j.jbmt.2016.06.001. Epub 2016 Jun 11. PMID 28167167
- [Background] Taimur M, Shah MAA, Ali M, Barry HD, Hussain SZM, Shahzad H, Rizwan A. Frequency of Cognitive Impairment in Patients with Parkinson's Disease. Cureus. 2019 May 23;11(5):e4733. doi: 10.7759/cureus.4733. PMID 31355092
- [Background] Yuan RY, Chen SC, Peng CW, Lin YN, Chang YT, Lai CH. Effects of interactive video-game-based exercise on balance in older adults with mild-to-moderate Parkinson's disease. J Neuroeng Rehabil. 2020 Jul 13;17(1):91. doi: 10.1186/s12984-020-00725-y. PMID 32660512
- [Background] Santos P, Machado T, Santos L, Ribeiro N, Melo A. Efficacy of the Nintendo Wii combination with Conventional Exercises in the rehabilitation of individuals with Parkinson's disease: A randomized clinical trial. NeuroRehabilitation. 2019;45(2):255-263. doi: 10.3233/NRE-192771. PMID 31498138
- [Background] Cabrera-Martos I, Jimenez-Martin AT, Lopez-Lopez L, Rodriguez-Torres J, Ortiz-Rubio A, Valenza MC. Effects of a core stabilization training program on balance ability in persons with Parkinson's disease: a randomized controlled trial. Clin Rehabil. 2020 Jun;34(6):764-772. doi: 10.1177/0269215520918631. Epub 2020 Apr 29. PMID 32349543